CLINICAL TRIAL: NCT03373591
Title: Randomized Controlled Trial Investigating Use of Liposomal Bupivacaine in Bariatric Surgery
Brief Title: Liposomal Bupivacaine in Bariatric Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Diego Camacho, Director Minimally Invasive and Endoscopic Surgery, Fellowship Program Director, Associate Professor of Surgery Albert Einstein College of Medicine, Montefiore Medical Center, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-7706
Record Dates: First submitted 2017-12-09; First posted 2017-12-14 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Bariatric Surgery Analgesia
Keywords: bariatric surgery; liposomal bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Liposomal Bupivacaine TAP block (Experimental): Patients will be randomized to receive an intraoperative transverse abdominis peritoneal (TAP) block with liposomal bupivacaine (LB). The solution used to perform the TAP block with LB will comprise of 20mL of liposomal bupivacaine solution, 30mL of 0.25% bupivacaine, and 100mL of normal saline.
  Interventions: Drug: Liposomal Bupivacaine TAP block
- Regular Bupivacaine TAP block (Active Comparator): Patients will be randomized to receive an intraoperative transverse abdominis peritoneal (TAP) block with regular bupivacaine (RB).The solution used to perform the TAP block with RB will comprise of 50mL of 0.25% bupivacaine and 100mL of normal saline.
  Interventions: Drug: Bupivacaine TAP block
- No TAP block (No Intervention): Patients will be randomized to receive no TAP block as a control group.

INTERVENTIONS:
Drug: Liposomal Bupivacaine TAP block — Infiltration of the transverse abdominis peritoneum by a local anesthetic under laparoscopic visualization.
  Other Names: Exparel TAP block
  Arms: Liposomal Bupivacaine TAP block
Drug: Bupivacaine TAP block — Infiltration of the transverse abdominis peritoneum by a local anesthetic under laparoscopic visualization.
  Arms: Regular Bupivacaine TAP block

SUMMARY:
The aim of this study is to perform a randomized controlled trial for patients undergoing bariatric surgery, comparing the need for opiates with and without administration of a transversus abdominis plane (TAP) block using the long acting local anesthetic, liposomal bupivacaine (Exparel®). From this study, the investigators will assess whether use of long acting local anesthetic can reduce the need for opiates in the bariatric population.

DETAILED DESCRIPTION:
A prospective randomized controlled trial investigating the use of long acting local anesthetic for transversus abdominis block in patients undergoing bariatric surgery at Montefiore Medical Center. Patients will be randomized to either receive an intraoperative TAP block with LB, an intraoperative TAP block with RB, or no TAP block. All participants will receive standard post-operative analgesia regimen. Pain scores will be recorded by the nursing staff as reported by the patients for 24-36 hours post surgery. Patients will be monitored for secondary post-operative complications up to the 2-week mark following intervention.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients undergoing bariatric surgery (LSG or LRYGB)
* Patients 18 years of age and older
* Surgical treatment between 01/01/2018 and 12/31/2018 over a 1 year period

Exclusion Criteria:

* Patients under the age of 18 years old
* Patients taking any opiates within 30 days of enrollment in the trial
* Patients with a history of chronic pain.
* Patients taking pregabalin or gabapentin.
* ASA IV
* Prior laparotomy
* Body Mass Index ≥ 60 kg/m2
* History of cardiac arrhythmia
* History of Seizure
* Psychiatric Diagnosis currently on antipsychotic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine TAP Block: Patients were randomized to receive an intraoperative transverse abdominis peritoneal (TAP) block with liposomal bupivacaine (LB). The solution used to perform the TAP block with LB was composed of 20mL of liposomal bupivacaine solution, 30mL of 0.25% bupivacaine, and 100mL of normal saline.
  Liposomal Bupivacaine TAP block: Infiltration of the transverse abdominis peritoneum by a local anesthetic under laparoscopic visualization.
- Regular Bupivacaine TAP Block: Patients were randomized to receive an intraoperative transverse abdominis peritoneal (TAP) block with regular bupivacaine (RB).The solution used to perform the TAP block with RB was composed of 50mL of 0.25% bupivacaine and 100mL of normal saline.
  Bupivacaine TAP block: Infiltration of the transverse abdominis peritoneum by a local anesthetic under laparoscopic visualization.
- No TAP Block: Patients were randomized to receive no TAP block as a control group.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Started | 75 | 71 | 73
Completed | 75 | 71 | 73
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block | Total
Number analyzed (Participants) | 75 | 71 | 73 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (9.8) | 39.4 (10.9) | 40.4 (11.0) | 40.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 55 | 66 | 181
  Male | 15 | 16 | 7 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 26 | 25 | 76
  White | 16 | 4 | 7 | 27
  More than one race | 34 | 40 | 39 | 113
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 75 | 71 | 73 | 219
Weight [Mean (Standard Deviation); unit: Kilograms] | 119.5 (23.8) | 121.7 (22.6) | 116.6 (20.2) | 119.3 (22.2)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 44.5 (7.6) | 44.8 (5.5) | 44.2 (5.5) | 44.5 (6.2)
Procedure [Count of Participants; unit: Participants]
  Gastric Bypass | 15 | 16 | 21 | 52
  Sleeve Gastrectomy | 55 | 55 | 50 | 160
  Sleeve to Bypass Conversion | 5 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Fentanyl PCA mcg
Description: Fentanyl PCA (patient controlled analgesia) total microgram usage.
Time Frame: 24 hours post surgery.
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Micrograms | 351.4 (209.4) | 360.7 (223.5) | 353.9 (231.0)

2. Primary Outcome: Total Fentanyl Usage
Description: Total fentanyl usage in micrograms, including both PCA and IV push administered medication.
Time Frame: During hospitalization, up to 7 days.
Measure: Mean (Standard Deviation); unit: Micrograms
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Micrograms | 424.1 (222.9) | 434.2 (237.4) | 427.5 (245.8)

3. Secondary Outcome: Acetaminophen Usage
Description: Total amount of acetaminophen used for analgesia.
Time Frame: During hospitalization, up t 7 days.
Measure: Mean (Standard Deviation); unit: Miligrams
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Miligrams | 486.4 (553.1) | 501.0 (456.0) | 353.4 (486.9)

4. Secondary Outcome: NSAID Usage
Description: Total amount of NSAID (ketorolac) use for analgesia.
Time Frame: During hospitalization, up to 7 days.
Measure: Mean (Standard Deviation); unit: Miligrams
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Miligrams | 14.2 (30.2) | 42.5 (21.5) | 21.3 (30.5)

5. Secondary Outcome: Pain Score
Description: Patient reported composite measure pain score, with a total range of 0 to 10, with 0 being the absence of pain, 1 being the least amount of pain and 10 being the highest amount of pain.
Time Frame: 24 hours post surgery.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
units on a scale | 4.3 (1.7) | 4.7 (1.7) | 4.7 (1.5)

6. Secondary Outcome: Length of Stay
Description: Hours of hospitalization post-surgery
Time Frame: Assessed every 24 hours post surgery, up to 168 hour post-surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Participants
  24 hours | 42 | 44 | 46
  48 hours | 26 | 26 | 25
  72 hours | 5 | 1 | 1
  96 hours | 1 | 0 | 0
  120 hours | 1 | 0 | 0
  168 hours | 0 | 0 | 1

7. Secondary Outcome: Nausea
Description: Number of participants with presence or absence of nausea reported and recorded by the nurse.
Time Frame: 24 hours post surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Participants | 27 | 41 | 34

8. Secondary Outcome: Time to Ambulation
Time Frame: Assessed every 24 hours post surgery, up to 168 hour post-surgery.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
Number analyzed (Participants) | 75 | 71 | 73
Hours | 51 (1.7) | 60 (1.6) | 59 (2.0)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks post-procedure.
Arm/Group | Liposomal Bupivacaine TAP Block | Regular Bupivacaine TAP Block | No TAP Block
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/71 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/71 | 0/73
Other Adverse Events (participants affected / at risk) | 0/75 | 0/71 | 0/73

LIMITATIONS AND CAVEATS:
Further studies are needed to attempt to match patients based on variables that effect opiate metabolism and pain response, and to include alternative secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT03373591/Prot_SAP_000.pdf